CLINICAL TRIAL: NCT02508259
Title: The UCSD Suramin Autism Treatment-1 (SAT1) Trial
Brief Title: University of California, San Diego (UCSD) Suramin Autism Treatment-1 (SAT1) Trial
Acronym: SAT1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Robert K. Naviaux, Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-0134
Record Dates: First submitted 2015-07-22; First posted 2015-07-24 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Autism Spectrum Disorders
Keywords: mitochondria; purinergic signaling; cell danger response
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Suramin; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Suramin (Active Comparator): 20 mg/kg suramin in 50 ml of saline by intravenous infusion over 30 minutes
  Interventions: Drug: Suramin
- Saline (Placebo Comparator): 50 ml of saline by intravenous infusion over 30 minutes
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Suramin — 20 mg/kg IV in 50 ml saline over 30 minutes
  Other Names: Germanin
  Arms: Suramin
Drug: Saline — 50 ml IV over 30 minutes
  Other Names: Normal saline
  Arms: Saline

SUMMARY:
This study is designed to test the safety and efficacy of a single, intravenous dose of suramin in autism spectrum disorders (ASD).

DETAILED DESCRIPTION:
This study is designed to test a new theory of the origin and treatment of ASD. In this theory, ASD is caused by both genes and environment interacting to produce a persistent cell danger response (CDR; Naviaux RK, 2014) that interferes with and alters normal child brain development. Gut microbiome and immune systems are also affected. In this theory, the pathological persistence of the cell danger response is traceable to mitochondria, and maintained by purinergic signaling mediated by the release of extracellular nucleotides like adenosine triphosphate (ATP), adenosine diphosphate (ADP), uridine triphosphate (UTP), and uridine diphosphate (UDP). Suramin inhibits excess purinergic signaling by acting as a competitive inhibitor of nucleotide signaling at both ionotropic purinergic (P2X) receptors, and G-protein coupled, metabotropic purinergic (P2Y) receptors. Suramin has been found to correct the symptoms, metabolism, and brain synaptic abnormalities in two classical genetic and environmental mouse models of autism (Naviaux JC, et al. 2015; Naviaux JC, et al. 2014; Naviaux RK, et al. 2013). This study will test the safety and efficacy of a single dose of suramin in children with ASD. While it is not anticipated that a single dose will produce benefits for more than a few weeks, if successful, this study may lead to the development of newer and safer drugs for autism treatment.

ELIGIBILITY:
Inclusion Criteria:

* Autism diagnostic observation schedule (ADOS) score of ≥ 7
* Diagnosis of autism spectrum disorder by Diagnostic and Statistical Manual, 5th edition (DSM-V)
* Stable treatment and diet regimen for ≥ 2 months
* Resident of San Diego region

Exclusion Criteria:

* Any prescription medications
* Hospitalization within the previous 2 months
* Active medical problem such as seizures, heart, liver, kidney, or adrenal disease
* Planning to start a new drug, diet, or behavioral intervention during the study
* Weight under the 5th percentile for age
* Unable to tolerate venipuncture, urine collection, or an indwelling intravenous catheter for 3-4 hours
* Plasma creatinine ≥ 1.4 mg/dl
* Liver function alanine amino transferase (ALT) or aspartate amino transferase (AST) ≥ 1.5-fold above the upper limit of normal
* Known intolerance to suramin or other antipurinergic drugs
* Unable to perform or cooperate with study requirements

Ages: 4 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert K Naviaux, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego School of Medicine, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Safety, metabolomic, and completed outcome data will be made available to qualified institutional groups after peer review and publication.

REFERENCES:
- [Background] Naviaux JC, Wang L, Li K, Bright AT, Alaynick WA, Williams KR, Powell SB, Naviaux RK. Antipurinergic therapy corrects the autism-like features in the Fragile X (Fmr1 knockout) mouse model. Mol Autism. 2015 Jan 13;6:1. doi: 10.1186/2040-2392-6-1. eCollection 2015. PMID 25705365
- [Background] Naviaux JC, Schuchbauer MA, Li K, Wang L, Risbrough VB, Powell SB, Naviaux RK. Reversal of autism-like behaviors and metabolism in adult mice with single-dose antipurinergic therapy. Transl Psychiatry. 2014 Jun 17;4(6):e400. doi: 10.1038/tp.2014.33. PMID 24937094
- [Background] Naviaux RK, Zolkipli Z, Wang L, Nakayama T, Naviaux JC, Le TP, Schuchbauer MA, Rogac M, Tang Q, Dugan LL, Powell SB. Antipurinergic therapy corrects the autism-like features in the poly(IC) mouse model. PLoS One. 2013;8(3):e57380. doi: 10.1371/journal.pone.0057380. Epub 2013 Mar 13. PMID 23516405
- [Background] Naviaux RK. Metabolic features of the cell danger response. Mitochondrion. 2014 May;16:7-17. doi: 10.1016/j.mito.2013.08.006. Epub 2013 Aug 24. PMID 23981537
- [Background] Naviaux RK, Curtis B, Li K, Naviaux JC, Bright AT, Reiner GE, Westerfield M, Goh S, Alaynick WA, Wang L, Capparelli EV, Adams C, Sun J, Jain S, He F, Arellano DA, Mash LE, Chukoskie L, Lincoln A, Townsend J. Low-dose suramin in autism spectrum disorder: a small, phase I/II, randomized clinical trial. Ann Clin Transl Neurol. 2017 May 26;4(7):491-505. doi: 10.1002/acn3.424. eCollection 2017 Jul. PMID 28695149
- See also: Resource materials from the PI's lab website — http://naviauxlab.ucsd.edu/science-item/autism-research/

RESULTS

PARTICIPANT FLOW:
Groups:
- Suramin: 20 mg/kg IV x1
- Saline (Placebo): IV Infusion x 1
Period: Overall Study
Arm/Group | Suramin | Saline (Placebo)
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Male subjects with autism spectrum disorder (ASD), ages 4-17 years
Groups:
- Suramin: 20 mg/kg IV x 1
- Total: Total of all reporting groups
Arm/Group | Suramin | Saline (Placebo) | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.9 (3.3) | 9.2 (3.8) | 9.1 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Autism Diagnostic Observation Schedule, 2nd edition (ADOS2) [Mean (Standard Deviation); unit: units on a scale] — ADOS2 comparison scores are units on a scale of 0-10. A score of 7-10 was required for enrollment. A score of 7-10 is diagnostic for autism spectrum disorder (ASD). The higher the score, the more severe the core symptoms of autism spectrum disorder. Scores of 6 and below are considered off the ASD spectrum.
  units on a scale | 8.6 (0.9) | 9.4 (1.3) | 9.0 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Autism Diagnostic Observation Schedule, 2nd Edition (ADOS2)
Description: ADOS2 comparison scores are units on a scale of 0-10. A score of 7-10 was required for enrollment. A score of 7-10 is diagnostic for autism spectrum disorder (ASD). The higher the score, the more severe the core symptoms of autism spectrum disorder. Scores of 6 and below are considered off the ASD spectrum.
Time Frame: 6 weeks compared to baseline
Population: Patients receiving either suramin or saline.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Saline (Placebo): IV Infusion
Arm/Group | Suramin | Saline (Placebo)
Number analyzed (Participants) | 5 | 5
units on a scale | -1.6 (0.55) | -0.4 (0.55)
Statistical Analysis 1: Comparison: Suramin; In this analysis, each child was used as their own control to examine before and after suramin treatment effects in a paired t-test design. This study was a small pilot study of safety and activity of suramin. The small subject numbers of just 5 per group make it impossible to draw any strong conclusions about efficacy. Future studies are required; Test type: Equivalence — The null hypothesis was that before and after treatment ADOS scores were equivalent; p = 0.0028, t-test, 2 sided; Mean Difference (Net) = -1.6, 95% CI 2-sided [-2.3 to -0.9], Standard Deviation 0.55

2. Primary Outcome: Expressive Language
Description: Expressive One Word Picture Vocabulary Test (EOWPVT) scores are normalized for age. Typical language development produces a mean score of 100 with a standard deviation of 15. Outcomes for EOWPVT were expressed as the mean of the child-specific difference before and 6-weeks after treatment. For example, if the 6-week standard EOWPVT score was 59.6 and the baseline score was 63.8, the difference is -4.2 (= 59.6 - 63.8). A decrease in score at 6 weeks would corresponds to a decrease in language performance, while an increase, a positive difference, would reflect an increase.
Time Frame: 6 weeks compared to baseline
Population: Subjects receiving either suramin or saline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Suramin | Saline (Placebo)
Number analyzed (Participants) | 5 | 5
units on a scale | -4.2 (8.3) | 2.0 (4.6)
Statistical Analysis 1: Comparison: Suramin; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — The child-specific difference in EOWPVT scores were compared for equivalence before and 6-weeks after suramin treatment; p = 0.32, t-test, 2 sided; Mean Difference (Net) = -4.2, 95% CI 2-sided [-14.5 to 6.1], Standard Deviation 8.3

3. Secondary Outcome: Aberrant Behavior Checklist (ABC)
Description: The full ABC is a 58-item parent rating with five factors: Irritability, Social Withdrawal, Stereotypy, Hyperactivity and Inappropriate Speech. Stereotypy is reported, and scores range from 0 to 21, with higher scores indicating worse behavior. A negative difference corresponds to decreased symptoms after treatment. A positive difference corresponds to increased symptoms after treatment.
Time Frame: 6 weeks compared to baseline
Population: Subjects receiving either suramin or saline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Suramin | Saline (Placebo)
Number analyzed (Participants) | 5 | 5
units on a scale | -4.0 (2.3) | 1.0 (4.3)
Statistical Analysis 1: Comparison: Suramin; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — In this analysis, the null hypothesis was tested that the child-specific ABC subscores for stereotypy were unchanged before and after suramin treatment; p = 0.019, t-test, 2 sided; Mean Difference (Net) = -4.0, 95% CI 2-sided [-6.9 to -1.1], Standard Deviation 2.3

4. Secondary Outcome: Autism Treatment Evaluation Checklist (ATEC)
Description: The reported value is the Language sub-score of the ATEC, and the range for the language sub-score is 0-20. The higher the score, the worse the disability. Outcomes were measured at 6 weeks after treatment compared to baseline. A negative difference corresponds to a decrease in language disability, i.e an improvement in speech and language. A positive difference reflects an increase in language disability, i.e. a decrease in speech and language.
Time Frame: 6 weeks
Population: Subjects receiving either suramin or saline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Suramin | Saline (Placebo)
Number analyzed (Participants) | 5 | 5
units on a scale | -2.0 (1.4) | -0.2 (2.9)
Statistical Analysis 1: Comparison: Suramin; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — In this analysis, we tested the equivalence of the child-specific ATEC subscore for language before and 6-weeks after treatment with suramin; p = 0.034, t-test, 2 sided; Mean Difference (Net) = -2.0, 95% CI 2-sided [-2.7 to -0.49], Standard Deviation 1.4

5. Secondary Outcome: The Clinical Global Impression - Improvement Scale (CGI-I)
Description: The CGI-I is scale that ranges from 1-7, reflecting the change in core autism behaviors after treatment. 1 is much improved, 4 is unchanged, and 7 is much worse.
Time Frame: Overall ASD symptoms at 6 weeks
Population: Subjects receiving either suramin or saline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Suramin | Saline (Placebo)
Number analyzed (Participants) | 5 | 5
units on a scale | -1.8 (1.04) | 0.0 (0.34)
Statistical Analysis 1: Comparison: Suramin vs Saline (Placebo); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — In this analysis, overall ASD symptom scores, measured by CGI were compared between suramin and placebo groups; p = 0.05, ANOVA; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-3.4 to -0.15], Standard Deviation 1.04

6. Secondary Outcome: Repetitive Behavior Questionnaire
Description: Total repetitive behavior was assessed using the Repetitive behavior questionnaire (RBQ), which has a scale from 0-87. Higher scores correspond to more severe repetitive behavior. Outcomes were analyzed as the difference in the score 6 weeks after treatment compared to baseline. A negative difference corresponds to improved behavior compared to baseline. A positive difference corresponds to worse behavior.
Time Frame: 6 weeks compared to baseline
Population: Subjects receiving suramin or saline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Suramin | Saline (Placebo)
Number analyzed (Participants) | 5 | 5
units on a scale | -3.2 (5.8) | -0.8 (3.3)
Statistical Analysis 1: Comparison: Suramin; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — In this analysis, the child-specific RBQ score was tested for equivalence before and 6-weeks after suramin treatment; p = 0.28, t-test, 2 sided; Mean Difference (Net) = -3.2, 95% CI 2-sided [-10.4 to 4.0], Standard Deviation 5.8

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Suramin | Saline (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suramin (N=5) | Saline (Placebo) (N=5)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Upper respiratory tract infection (URI) (Infections and infestations) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) — In 7-year old after pizza and slushee consumption after playing youth league basketball, and in a 6-year old after a car ride.
Hyperactivity (Nervous system disorders) | 2 (2) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) — Both cases occurred 6-weeks after the infusion, after several days of a URI and fasting before lunch for the blood draw. Hypoglycemia was asymptomatic and corrected after a normal lunch.
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No